CLINICAL TRIAL: NCT00405080
Title: An Open-Label, Two Period, Fixed Sequence Study of Healthy Subjects to Assess the Effect of Repeat Oral Dosing of [Rifampin] on the Pharmacokinetics of a Single Oral Dose of [GW679769]
Brief Title: A Study in Healthy Subjects to Assess How Dosing of Rifampin Affects What the Body Does to a Dose of GW679769 (Casopitant).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKV105091
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Nausea and Vomiting, Chemotherapy-Induced
Keywords: Rifampin GW679769
MeSH Terms: conditions — Nausea; Vomiting | interventions — casopitant; Rifampin

ARMS (2):
- Treatment Period 1 (Experimental): Subject will receive single oral dose of 150 milligram (mg) of Casopitant. There will be wash out period of 7 days.
  Interventions: Drug: GW679769 (Casopitant) oral tablets
- Treatment Period 2 (Experimental): Subjects will receive rifampin 600 mg once daily on Days 1 - 9. On Day 8 subjects will receive a single dose of oral casopitant 150 mg along with rifampin.
  Interventions: Drug: GW679769 (Casopitant) oral tablets; Drug: Rifampin oral capsules

INTERVENTIONS:
Drug: GW679769 (Casopitant) oral tablets — Casopitant tablets will be available with dose strength of 50 mg. Subjects will receive three 50 mg tablets for the dose of 150 mg. On Day 8 of Treatment Period 2, the dose of casopitant and rifampin is to be taken at the same time.
Drug: Rifampin oral capsules — Rifampin capsules will be available with dose strength of 300 mg. Subjects will receive two 300 mg capsules for the dose of 600 mg. On Day 8 of Treatment Period 2, the dose of casopitant and rifampin is to be taken at the same time.
  Other Names: GW679769 (Casopitant) oral tablets
  Arms: Treatment Period 2

SUMMARY:
This study will examine what the body does while taking GW679769 alone and together with rifampin in healthy adult subjects.

ELIGIBILITY:
Inclusion criteria:

* healthy
* female subjects who cannot become pregnant
* able to swallow and keep down oral medication
* can understand and follow the protocol requirements and instructions

Exclusion criteria:

* smokes at least 4 packs per day in the past 12 months
* use of prescription or non-prescription drug(s)
* herbal or dietary supplements or vitamins with 14 days prior to first dose of study medication
* a clinically relevant abnormality medical condition or circumstance making the subject unsuitable for the study per the study doctor
* blood donation in excess of 1 pint within 56 days before dosing of medication
* iron deficient
* history or drug allergy of study medication
* history of drug or alcohol abuse or dependency within the past 6 months
* subjects cannot use any nicotine-containing products within the last 6 months
* positive for HIV, Hepatitis B or C
* active peptic ulcer disease
* uncontrolled nausea and vomiting
* active infection
* heart failure
* female who is lactating
* female who has a positive pregnancy test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-11-11 (Actual); Primary Completion 2007-01-05 (Actual); Study Completion 2007-01-05 (Actual)

PRIMARY OUTCOMES:
Plasma levels for casopitant will be measured in Period 1 at Day 1 to 3 and in Period 2 at Day 8. Plasma levels for rifampin will be measured in Period 2 at Day 8 to 10. | Up to Day 10

SECONDARY OUTCOMES:
clinical lab tests adverse events vital signs 12 lead ECGs liver function tests | Up to Day 12

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study NKV105091 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/NKV105091?search=study&search_terms=NKV105091#rs
- Available data/document: Clinical Study Report: NKV105091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: NKV105091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKV105091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: NKV105091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKV105091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: NKV105091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register